CLINICAL TRIAL: NCT05215509
Title: Exercise-induced Cardiac Adaptions in Rheumatoid Arthritis Patients During Interleukin-6 vs. Tumor Necrosis Factor Antibody Therapy: a Randomised, Controlled Study.
Brief Title: Exercise-induced Cardiac Adaptions in Rheumatoid Arthritis Patients During IL-6 vs. TNF Antibody Therapy
Acronym: RABEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Regitse Christensen, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-21010559
Record Dates: First submitted 2021-11-16; First posted 2022-01-31 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Cardiac adaptations; Metabolic adaptations; High intensity interval training
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Exercise; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RA patients TNFi Exercise (Experimental): The patients will be randomized to 12-week supervised exercise training intervention or no exercise training. The exercise training program includes three supervised sessions per week over a 12-week period.
  The program consists of high intensity endurance training on ergometer bicycles. The intensity will progress throughout the 12 weeks of training. The training consists of 10 minutes of warm up at 40-60% maximum heart rate (HRmax), followed by 25 minutes of high intensity interval training (4 bouts of 4 min at >85% HRmax interspaced by 3 minutes of low intensity training at 40-60% Hrmax) and finally a 5 min cool-down of 50% Hrmax
  Interventions: Behavioral: Exercise
- RA patients TNFi Control (Active Comparator): This group will be allocated to "control" and therefore no supervised exercise regimen
  Interventions: Behavioral: No exercise
- RA patients IL-6Rb Exercise (Experimental): The patients will be randomized to 12-week supervised exercise training intervention or no exercise training. The exercise training program includes three supervised sessions per week over a 12-week period.
  The program consists of high intensity endurance training on ergometer bicycles. The intensity will progress throughout the 12 weeks of training. The training consists of 10 minutes of warm up at 40-60% maximum heart rate (HRmax), followed by 25 minutes of high intensity interval training (4 bouts of 4 min at >85% HRmax interspaced by 3 minutes of low intensity training at 40-60% Hrmax) and finally a 5 min cool-down of 50% Hrmax
  Interventions: Behavioral: Exercise
- RA patients IL-6Rb Control (Active Comparator): This group will be allocated to "control" and therefore no supervised exercise regimen
  Interventions: Behavioral: No exercise

INTERVENTIONS:
Behavioral: Exercise — Supervised high-intensity interval training for 12 weeks three times per week. The supervision may be physical or online supervision
  Other Names: High intensity interval training
  Arms: RA patients IL-6Rb Exercise; RA patients TNFi Exercise
Behavioral: No exercise — Control group, therefore no supervised exercise regime
  Arms: RA patients IL-6Rb Control; RA patients TNFi Control

SUMMARY:
The present study will investigative the physiological effects of the cytokines interleukin-6 (IL-6) and tumor necrosis factor (TNF) on the adaptive changes to exercise in patients with rheumatoid arthritis. The investigators hypothesize that blockage of IL-6 receptors will decrease the cardiac and metabolic adaptations to exercise training compared to the inhibition of TNF. 80 patients will be included in a 12-week investigator blinded randomised exercise training intervention study.

DETAILED DESCRIPTION:
80 patients with rheumatoid arthritis who are being treated with either interleukin-6 receptor blockers (IL-6Rb) or tumor necrosis factor inhibitors (TNFi) for a minimum of four months prior to enrollment will be recruited and undergo baseline testing, including examination, biochemistry, ECG, DXA, OGTT, pulmonary function, VO2max, echocardiography, cardiac MRI.

After baseline testing, 40 patients in IL-6 receptor blocker treatment and 40 patients in TNF inhibitor treatment.will be randomly allocated into one group receiving standard of care (control group) or a group performing supervised high-intensity interval training three times a week over a period of 12 weeks. The randomization procedure involves a computer-generated block randomization schedule in a ratio of 1:1 stratified by sex by an independent person. Following the 12-week intervention period, all groups will complete a series of follow-up tests (as baseline testing).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 and <70 years
* Informed consent
* Diagnosed RA based on the 2010 American College of Rheumatology/ EULAR criteria. In biological treatment with either IL-6rB og TNFi over four months prior to enrollment
* Low RA disease activity, based on the Disease Activity Score-28 ESR for Rheumatoid Arthritis (DAS28) <=3.2
* An electrocardiogram without features of left ventricular hypertrophy defined by the European Society of Cardiology
* Females of childbearing potential have to use one or more of the following highly effective methods for contraception in order to be included:

  * Vasectomized partner
  * Bilateral tubal occlusion
  * Sexual abstinence
  * Intrauterine device
  * Hormonal contraception
* Females who are considered to have no childbearing potential are

  * Bilateral tubal ligation
  * Bilateral oophorectomy
  * Complete hysterectomy
  * Postmenopausal defined as 12 months with no menses without an alternative medical cause

Exclusion Criteria:

* Health conditions that prevent participating in the exercise intervention determined by the Project Coordinator
* Subjects who cannot undergo MRI scans (metallic implants or claustrophobia)
* Corticosteroid use per os > 10 mg/day within seven days of study enrollment
* Intramuscular corticosteroid within 3 weeks of the study enrollment
* Grade 2 hypertension (systolic BP > 160 mmHg and/or diastolic BP >100 mmHg) despite the use of antihypertensive drugs.
* Pregnancy
* Subjects with insulin dependent Diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular mass | 12 weeks
  measured by MRI scan

SECONDARY OUTCOMES:
Visceral adipose tissue mass | 12 weeks
  measured by MRI scan
Stroke volume | 12 weeks
  Structural cardiac parameter: measured by MRI scan and echocardiography
Left ventricular and atrial end-diastolic volume | 12 weeks
  Structural cardiac parameter: measured by MRI scan and echocardiography
LVEF | 12 weeks
  Functional cardiac parameters: measured by MRI scan and echocardiography
Global longitudinal strain | 12 weeks
  Functional cardiac parameters: measured by MRI scan and echocardiography
E/A ratio | 12 weeks
  Functional cardiac parameters: measured by MRI scan and echocardiography
E/é | 12 weeks
  Functional cardiac parameters: measured by MRI scan and echocardiography
Left ventricular and atrial end-systolic volume | 12 weeks
  Structural cardiac parameter: measured by MRI scan and echocardiography
Left atrial volume index | 12 weeks
  Structural cardiac parameter: measured by MRI scan and echocardiography
Interventricular septum thickness | 12 weeks
  Structural cardiac parameter: measured by MRI scan and echocardiography
Left ventricular posterior wall thickness | 12 weeks
  Structural cardiac parameter: measured by MRI scan and echocardiography
Aortic and pulmonary distensibility and pulse wave velocity | 12 weeks
  Functional vascular parameter: measured by MRI
Subcutaneous, visceral and epicardial adipose tissue | 12 weeks
  Measured by MRI and MR spectroscopy
Intramyocardial triglyceride content | 12 weeks
  Measured by MRI and MR spectroscopy
Cardiorespiratory fitness | 12 weeks
  Measured with an incremental VO2 protocol on exercise bike
Dynamic spirometry | 12 weeks
  Pulmonary function testing
Whole body plethysmography | 12 weeks
  Pulmonary function testing
Diffusion capacity | 12 weeks
  Pulmonary function testing
Body composition | 12 weeks
  Measured by a DXA scan
Oral glucose tolerance test | 12 weeks
  75g of glucose taken while fasting
Axial accelerometer-based physical activity monitors | 5 days in week 6 of the intervention/control
  Free-living physical activity is measured using axial accelerometer-based physical activity monitors (AX3; Axivity, Newcastle upon Tyne, UK) for a 5-day period
Dietary intake | 3 days in the week 6 of intervention/control
  Self reported intake of all foods and liquids
Blood sample | 12 weeks
  Change in fasting total cholesterol, low-density lipoprotein (LDL)-cholesterol and high-density lipoprotein (HDL)-cholesterol (mmol/L). Following an overnight fast (10 hours), blood samples are collected and processed by a trained laboratory technician and analysed according to standard procedures.
Blood sample | 12 weeks
  Change in triglycerides (mmol/L). Following an overnight fast (10 hours), blood samples are collected and processed by a trained laboratory technician and analysed according to standard procedures.
RA disease specific outcomes 1 | 12 weeks
  Change in measures of the international Core Outcome Set for rheumatoid arthritis : 66/68 tender and swollen joint count
RA disease specific outcomes 2 | 12 weeks
  Change in visual analogue scale (VAS) pain, VAS physician global assessment, VAS patient global assessment
  The Visual Analogue Scale (VAS) is a self-report measure consisting simply of a 100 mm horixontal line with a statement at each end representing one extreme (0mm = nothing, 100mm = extreme)
RA disease specific outcomes 3 | 12 weeks
  Change in Health Assessment Questionnaire (HAQ-DI)
  Total score is between 0-3.0. Increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment.
RA disease specific outcomes 4 | 12 weeks
  Change in Short Form 36 (SF-36) Health Survey Questionnaire
  A 8-scale score within 8 domains.All items are scored so that a high score defines a more favorable health state.
RA disease specific outcomes 5 | 12 weeks
  Change in the composite Disease Activity Score-28 ESR for Rheumatoid Arthritis (DAS28).
  A DAS28 of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission
RA disease specific outcomes 6 | 12 weeks
  Change in response criteria will be assessed according the clinical disease activity index (CDAI).
  The CDAI composite index quantifies disease activity in RA, by utilising four clinical parameters including tender and swollen joints and global assessment from both patient and assessor on a vasual analogue scale.
  CDAI interpretation score CDAI ≥ 22,1: High Activity CDAI < 22,1 og ≥10,1: Moderate Activity CDAI <10,0 og ≥ 2,9: Low Activity CDAI <2,9: Remission
RA disease specific outcomes 7 | 12 weeks
  Change in response criteria will be assessed according the American College of Rheumatology (ACR 20/50/70) response
RA disease specific outcomes 8 | 12 weeks
  Change in response criteria will be assessed according the European League Against Rheumatism (EULAR none/good/moderate response)

CONTACTS AND LOCATIONS:
Overall Officials: Regitse Christensen, Principal Investigator — Center for Physical Activity Research, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymised IPD obtained through this study may be provided to qualified researchers upon reasonable request.
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: Requests can be submitted following the publication of the primary outcome, and IPD will be accessible upon reasonable request up to 3 years from that date.
Access Criteria: Requests to acces IPD may be provided if a satisfactory research proposal is sent to Simon Jønck (simon.joenck.04@regionh.dk) and Regitse H Christensen (regitse.hoejgaard.Christensen@regionh.dk)

REFERENCES:
- [Derived] Jonck S, Adamsen ML, Rasmussen IE, Lytzen AA, Lok M, Vonsild Lund MA, Dreyer L, Jorgensen PG, Vejlstrup N, Kober L, Christensen R, Jacobsen S, Pedersen BK, Ellingsgaard H, Hojgaard P, Berg RMG, Christensen RH. IL-6 Inhibitors and TNF Inhibitors: Impact on Exercise-induced Cardiac Adaptations in Patients With Rheumatoid Arthritis. JACC Basic Transl Sci. 2025 May;10(5):551-563. doi: 10.1016/j.jacbts.2024.11.010. Epub 2025 Feb 5. PMID 40436519
- [Derived] Jonck S, Adamsen ML, Hojgaard P, Rasmussen IE, Ellingsgaard H, Lund MAV, Jorgensen PG, Jacobsen S, Kober L, Vejlstrup N, Dreyer L, Pedersen BK, Berg RMG, Christensen RH. Effect of a 12-week high-intensity exercise intervention: a comparison of cardiac exercise adaptations during biological disease-modifying antirheumatic drug treatment (TNF inhibitors vs IL-6 signalling inhibitors) in patients with rheumatoid arthritis - study protocol for a randomised controlled trial. BMJ Open. 2023 May 11;13(5):e068600. doi: 10.1136/bmjopen-2022-068600. PMID 37169504

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT05215509/SAP_000.pdf